CLINICAL TRIAL: NCT00487760
Title: African American Families and Lung Cancer Study
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907161; 07-HG-N161
Record Dates: First submitted 2007-06-16; First posted 2007-06-19 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-08-02

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; African-American Families; Genetic Risk Communication; Interest in Genetic Testing and Genetics Research; Health Disparities; Smoking Cessation
MeSH Terms: conditions — Lung Neoplasms; Smoking Cessation

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will learn more about the beliefs of family members of African American patients with lung cancer and whether these beliefs are associated with their interest in genetic testing for disease risk and willingness to participate in genetics research. Lung cancer is the second most common form of cancer and the leading cause of cancer deaths for men and women in the United States. Like most cancers, there are racial and ethnic disparities (gaps) in lung cancer cases and deaths. The age-adjusted rates for blacks and whites (years 2000 to 2003) was 76.9 per 100,000 and 66.0 per 100,000, respectively. Mortality rates were 62.5 per 100,000 for blacks and 55.3 per 100,000 for whites. Cigarette smoking is the most preventable cause of lung cancer. Findings are that African Americans begin smoking at older ages and smoke fewer cigarettes per day than Caucasian Americans do. Yet the severity of lung cancer is greater for African Americans. Behavioral, social, environmental, and genetic factors may explain the differences.

Participants (subjects) ages 18 to 55 who are family of patients with lung cancer who self-identify as African Americans may be eligible for this study. Washington, D.C., researchers plan to recruit 115 lung cancer patients and 200 family members-100 current smokers and 100 who never smoked. Lung cancer patients, who must have been born in the United States, will be recruited from those who are receiving care at the Washington Cancer Institute at the Washington Hospital Center. They will be asked to list relatives and friends they consider to be as close as family. Patients will be asked permission for researchers to contact those people. Family members will receive a letter telling them that unless they decline to participate, they will be contacted by a telephone interviewer.

The survey will feature questions to evaluate family members' explanations for the causes of lung cancer, as well as their reactions to possible reasons for the disparity in lung cancer between African Americans and Caucasian Americans. Subjects will be asked about perceived personal risk, worry about developing lung cancer, smoking history, motivation to quit smoking, feelings about the lung cancer patient's diagnosis, racial identify, experience with racial discrimination, pros and cons of genetic testing, and interest in genetic testing. The survey will take up to 20 minutes to complete.

This study may or may not have a direct benefit for those who participate. However, lung cancer patients and their families will be offered a free self-help guide to stop smoking. They will be referred to local smoking cessation programs. Knowledge gained from the study may be used to design smoking cessation methods and research studies related to genetics for minority populations.

DETAILED DESCRIPTION:
The purpose of the African American (AA) Families and Lung Cancer Study is to learn more about (1) the beliefs of family members of AA patients with lung cancer about why AA get lung cancer and (2) whether these beliefs are associated with their interest in genetic testing for lung cancer risk and willingness to participate in clinical genetics research. We plan to recruit 200 AAs (n = 100 current smokers and n = 100 never smokers) who are considered to be as close as family (both biological and non-biological kin) to patients with lung cancer who self-identify as AA (n = 115). Patients will be recruited from Washington Cancer Institute at the Washington Hospital Center in Washington, DC. Family members who self-identify as AA and are between the ages 18 and 55 will be eligible for the study. A Washington Hospital Center recruiter will approach patients and ask their willingness to be contacted for a telephone survey about their general well-being. As part of the survey, patients will be asked to enumerate family and friends who they consider to be as close as family, and asked to specifically focus on those who are current cigarette smokers and those who have never smoked. Patients will be asked to give permission to contact some or all of those enumerated. These family members will be mailed a letter to inform them that unless they call to decline they will be contacted by a telephone interviewer. The survey will include questions to assess family members' explanations for the causes of lung cancer and reactions to possible explanations for disparities in lung cancer between AA and Caucasian Americans (CA), perceived personal risk and worry about developing lung cancer, smoking history, motivation to quit smoking, emotional responses to the patient's diagnosis, racial identity, experience with racial discrimination, pros and cons of genetic testing, and interest in genetic testing (the primary outcome variable). Data analysis using hierarchical linear modeling will assess whether patient characteristics and family members' endorsement of genetics as the cause of lung cancer are associated with their interest in genetic testing and participation in clinical genetics research.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients:

In order to be included in this study, patients with lung cancer must meet inclusion criteria at 2 steps: (1) initial screening and written consent to be contacted by telephone, and (2) provision of verbal consent at the time of telephone contact to complete the survey.

Step 1a: In order to be approached about the study, patients must be (1) at least 18 years of age, (2) diagnosed with lung cancer at any stage (Stages Ia-IV), (3) approved for contact by their oncologist, and (4) identified by the recruiter or identified in medical records as Black.

Step 1b: In order to provide consent for contact for the telephone survey, patients must self-identify as AA/Black and must have been born in the U.S. Also, patients must be willing to give permission to contact at least one family member or friend considered as close as family who is a current cigarette smoker between the ages of 18 and 55 in order to provide consent.

Step 2: At the point of the patient survey, all patients will be asked their race/ethnicity. All patients who self-identify as AA/Black as defined by this research will be administered the patient survey.

Family:

Family members must self-identify as AA and be between the ages of 18 and 55 to be eligible for the study. Family also must meet the following inclusion criteria to be classified as either a current smoker (defined below) or a never smoker (defined below). These criteria for current smoker and never smoker are based on standard criteria used in smoking research.

Current Smoker: to be included as a smoker , the family member must report having smoked at least 100 cigarettes in their lifetime, and smoked 7 or more cigarettes in the past 7 days at the time of the family member survey.

Never Smokers: to be included as a never smoker , a family member must report no to having smoked at least 100 cigarettes in their lifetime.

EXCLUSION CRITERIA:

Former smokers (i.e., family who have smoked at least 100 cigarettes in their lifetime but smoked fewer than 7 cigarettes in the past 7 days) because previous research shows consistently that these individuals hold attitudes and beliefs more similar to those of current smokers than never smokers.

Patients who describe themselves as AA or Black but were not born in the U.S. will be excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-06-11; Study Completion 2011-08-02

CONTACTS AND LOCATIONS:
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Arthur CM, Katkin ES. Making a case for the examination of ethnicity of Blacks in United States Health Research. J Health Care Poor Underserved. 2006 Feb;17(1):25-36. doi: 10.1353/hpu.2006.0017. PMID 16520504
- [Background] Baty BJ, Kinney AY, Ellis SM. Developing culturally sensitive cancer genetics communication aids for African Americans. Am J Med Genet A. 2003 Apr 15;118A(2):146-55. doi: 10.1002/ajmg.a.10150. PMID 12655495
- [Background] Clark R, Anderson NB, Clark VR, Williams DR. Racism as a stressor for African Americans. A biopsychosocial model. Am Psychol. 1999 Oct;54(10):805-16. doi: 10.1037//0003-066x.54.10.805. PMID 10540593